CLINICAL TRIAL: NCT06389864
Title: High Frequency rTMS in Children and Adolescents With ADHD: a Randomized, Double Blind Clinical Trial.
Brief Title: rTMS in Children and Adolescents With ADHD:
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Salama Ahmed Omar, assistant lecturer at psychiatric department at assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rTMS in ADHD
Record Dates: First submitted 2024-04-02; First posted 2024-04-29 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: ADHD
Keywords: rTMS,ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real group (Active Comparator): rTMS administered at 10 Hz directed to the right dorsolateral prefrontal cortex. The pulse intensity was set at 80% of the observed motor threshold, 4 s on-train, 26 s off inter-train interval with 2000 pulses per session(29) for 5 sessions per week, for 15 sessions total (i.e., 30,000 pulses total in treatment course).
  Interventions: Device: rTMS (repetitive transcranial magnetic stimulation)
- Sham control group (Sham Comparator): the rTMS coil was tilted over the right dorsolateral pre-frontal cortex without touching the scalp administered at 10 Hz. The pulse intensity was set at 80% of the observed motor threshold, 4 s on-train, 26 s off inter-train interval with 2000 pulses per session for 5 sessions per week. for 15 sessions total.
  Interventions: Device: rTMS (repetitive transcranial magnetic stimulation)

INTERVENTIONS:
Device: rTMS (repetitive transcranial magnetic stimulation) — non invasive repetitive transcranial magnetic stimulation rTMS was administered at 10 Hz directed to the right dorsolateral prefrontal cortex. The pulse intensity was set at 80% of the observed motor threshold, 4 s on-train, 26 s off inter-train interval with 2000 pulses per session for 5 sessions per week, for 15 sessions total (i.e., 30,000 pulses total in treatment course) in the active TMS condition. For the sham rTMS, the coil was tilted over the right dorsolateral pre-frontal cortex without touching the scalp.

SUMMARY:
Assess the effect of RTMS on ADHD symptoms and assessment of this effect clinically and objectively.

DETAILED DESCRIPTION:
Sixty children with ADHD of both sexes and ages ranging between 8 and 16 years old were included in the study. Randomization of patients: Our patients in each subgroup were randomly allocated to intervention arms (real versus sham) by using serially numbered opaque closed envelopes. Each patient was placed in the appropriate group after opening the corresponding sealed envelope. The official sheet of the assiut university of Psychiatry was used for the assessment and interview. This includes demographic data, personal and family history, medical history, and mental state examination. All subjects were then assessed using the Full psychiatric interview (Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL) to diagnose ADHD and to exclude other diagnoses according to DSM5 classification, which took place in the first interview with the participants before the start of the study. An informed written consent was offered for the parents of the patients participating in the study. All participants were on drugs (stimulants and non-stimulants), and all other medications were stopped 2 weeks before the beginning of the study. Atomoxetine was (from 0.5 to 1.2 mg/ kg/day )(24-25-26) . thirty participants were allocated to the rTMS group who received 15 sessions of rTMS over the right DLPC, in conjunction with Atomoxetine 1.2 mg/kg/day. The other 30 participants were allocated to the Sham control group who received 15 sessions of sham rTMS and atomoxetine 1.2 mg/kg/day. All participants underwent assessments of the severity of ADHD symptoms done at 3 points, before the beginning of treatment (pre), after receiving 15 sessions of rTMS/Sham rTMS (post), and on follow-up 1 month after treatment (FU) (27), using Arabic version Conners' Parent Rating Scale - Revised Long form ,Clinical Global Impression and the resting motor threshold (RMT). The scores pre, post, and follow-up were compared to evaluate the improvement of clinical symptoms, and the therapeutic effects among the 2 groups were also compared. rTMS was delivered through a figure of 8 coil (the outer diameter of each wing is 9 cm, the maximum field strength=1.9 tesla) attached to a Magstim (UK) super rapid magnetic stimulator, (28) which administered at 10 Hz directed to the right dorsolateral prefrontal cortex, located at the F4 location from the EEG 10-20 system. The pulse intensity was set at 80% of the observed motor threshold, 4 s on-train, 26 s off inter-train interval with 2000 pulses per session(29) for 5 sessions per week, for 15 sessions total (i.e., 30,000 pulses total in treatment course) in the active TMS condition. For the sham rTMS, the coil was tilted over the right dorsolateral pre-frontal cortex without touching the scalp. Participants who received less than 75% of the number of sessions (12 sessions) were considered dropouts.

ELIGIBILITY:
Inclusion Criteria:

.Clinical diagnosis of ADHD met the diagnostic criteria for ADHD in the (DSM-5) of the American Psychiatric association.

.Must be able to swallow tablets.

.both sexes will be included in the study.

.Age will be 6-18 years.

.IQ≥70.

Exclusion Criteria:

* comorbid diagnosis of autism spectrum disorder, bipolar disorder, obsessive-compulsive disorder, conduct disorder, Tourette disorder or other tic disorders, schizophrenia, schizoaffective disorder, any other psychotic disorder or other.
* contraindications to magnetic stimulation such as any metallic object implanted in the skull (except for oral dental devices), an implanted medication pump or cochlear implant, implanted intra-cardiac lines or pacemaker.
* increase the risk of seizure with TMS such as a history of a seizure disorder, febrile seizures during childhood, known brain lesions, or a history of major head trauma involving loss of consciousness for more than 5 min were excluded from the study.
* major neurological deficits, disease, cerebral palsy other heart, liver, lung, kidney, or other serious somatic diseases.
* other medications or other treatment rather than treatment for ADHD. .Mood regulating medications within 14 days. .recent treatment with TMS.
* refuse to participate in the study or their caregiver refusing to give informed consent.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The resting motor threshold (RMT) | immediately after the end of sessions And follow up 1 month after the end sessions.
  was defined, according to the IFCN Committee recommendation, as the lowest stimulus intensity able to elicit MEPs of an amplitude >50 μV in at least 5 out of 10 trials, with the muscle at rest.
Arabic version Conners' Parent Rating Scale - Revised Long form | immediately after the end of sessions And follow up 1 month after the end sessions.
  is applied to detect the core symptoms of ADHD, detect its subtypes, and assess severity. It contains 80 items and can be completed by parents/guardians in approximately 20 minutes.
Clinical Global Impression CGI | immediately after the end of sessions And follow up 1 month after the end sessions.
  is designed to assess the effectiveness of a particular treatment: CGI-S assessing Illness Severity and CGI-C assessing Global Improvement or Change.

CONTACTS AND LOCATIONS:
Overall Officials: Yaser Mohamed Bader Elden elserogy, professor, Principal Investigator — processor at psychiatry department at assiut university hospital

REFERENCES:
- [Background] Thomas R, Sanders S, Doust J, Beller E, Glasziou P. Prevalence of attention-deficit/hyperactivity disorder: a systematic review and meta-analysis. Pediatrics. 2015 Apr;135(4):e994-1001. doi: 10.1542/peds.2014-3482. Epub 2015 Mar 2. PMID 25733754
- [Background] Biederman J, Spencer T, Wilens T. Evidence-based pharmacotherapy for attention-deficit hyperactivity disorder. Int J Neuropsychopharmacol. 2004 Mar;7(1):77-97. doi: 10.1017/S1461145703003973. Epub 2004 Jan 21. PMID 14733627
- [Background] Thapar A, Cooper M. Attention deficit hyperactivity disorder. Lancet. 2016 Mar 19;387(10024):1240-50. doi: 10.1016/S0140-6736(15)00238-X. Epub 2015 Sep 17. PMID 26386541
- [Background] Fitzgerald PB, Fountain S, Daskalakis ZJ. A comprehensive review of the effects of rTMS on motor cortical excitability and inhibition. Clin Neurophysiol. 2006 Dec;117(12):2584-96. doi: 10.1016/j.clinph.2006.06.712. Epub 2006 Aug 4. PMID 16890483
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Kumar G, Steer RA. Factorial validity of the Conners' Parent Rating Scale-revised: short form with psychiatric outpatients. J Pers Assess. 2003 Jun;80(3):252-9. doi: 10.1207/S15327752JPA8003_04. PMID 12763699
- [Background] Kujirai T, Caramia MD, Rothwell JC, Day BL, Thompson PD, Ferbert A, Wroe S, Asselman P, Marsden CD. Corticocortical inhibition in human motor cortex. J Physiol. 1993 Nov;471:501-19. doi: 10.1113/jphysiol.1993.sp019912. PMID 8120818